CLINICAL TRIAL: NCT04731155
Title: Impact of Early PCSK9 Inhibitor on Heart After Acute Myocardium
Brief Title: Impact of Early PCSK9 Inhibitor on Heart After Acute Myocardium Infarction
Acronym: PERFECT-AMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Hou Lei, Principal Investigator, Shanghai Tong Ren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021HL
Record Dates: First submitted 2021-01-23; First posted 2021-01-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Early PCSK9 Inhibitor on Ventricular Remodling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard group (Active Comparator)
  Interventions: Drug: standard medications
- experiment group (Experimental)
  Interventions: Drug: PCSK9 inhibitor （Alirocumab）plus standard medications

INTERVENTIONS:
Drug: PCSK9 inhibitor （Alirocumab）plus standard medications — PCSK9 inhibitor（Alirocumab） was giving to subjects before PPCI and continued twice a month until 3 month after AMI
  Arms: experiment group
Drug: standard medications — standard medications was giving to subjects according guidelines
  Arms: standard group

SUMMARY:
This is a prospect, multi-center, random study to investigate whether early offering PCSK9 inhibitor to acute myocardium infarction(AMI) can alleviate ventricular remodeling after primary percutaneous intervention(PPCI). Totally,twenty acute myocardium infarction subjects will be enrolled in this study after consent information. After randomization, the control group will receive standard therapy for AMI including PPCI. The experiment group will receive first PCSK9 inhibitor before PPCI, then twice a month until 3 months later. Six month after AMI, Myocardial salvage index will be used to evaluate ventricular remodeling. TnI peaking time and LDL control rates also will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age and less than 80 years old
2. Patients should have undergone successful percutaneous coronary intervention with drug-eluting stent for AMI and LAD should be the only culprit vessel.
3. Subject understand the study requirements and the treatment procedures and provided informed consent before the procedure

Exclusion Criteria:

1. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
2. Known hypersensitivity or contraindication to study medications
3. Plan to receive revascularization in next six month.
4. Have received revascularization before.
5. Subjects with life expectation less than one year.
6. Subjects with active malignant tumor
7. subjects with severe liver or renal dysfunction（ALT >5倍ULA，eGFR<15ml/min/1.73mm2）
8. Other conditions which the investigators think not applicable to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
myocardial salvage index measured by MRI | one week after PPCI
myocardial salvage index measured by MRI | six months after PPCI
eject fraction measured by MRI | one week after PPCI
eject fraction measured by MRI | six month after PPCI

SECONDARY OUTCOMES:
the change of serum level of TnI/T | 0,6 ,12,18 , 24 ,30,and 36 hours after PPCI
LDL -C control rate | the first month after PPCI
the serum lever of hsCRP | Baseline (before PPCI)
the serum lever of hsCRP | one week after PPCI

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongren Hospital, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai tenth people's hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No